CLINICAL TRIAL: NCT02496039
Title: A Study to Assess Effectiveness, Safety, and Health-related Outcomes of NUEDEXTA® (Dextromethorphan Hydrobromide and Quinidine Sulfate) for the Treatment of Pseudobulbar Affect (PBA) in Nursing Home Patients
Brief Title: Effectiveness, Safety, and Health-Related Outcomes of NUEDEXTA® in Nursing Home Patients With Pseudobulbar Affect (PBA)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated prematurely because of difficulty with recruiting.
Sponsor: Avanir Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15-AVR-404
Record Dates: First submitted 2015-07-08; First posted 2015-07-14 (Estimated); Results first posted 2017-07-03 (Actual); Last update posted 2017-07-03 (Actual); Status verified 2017-06

CONDITIONS: Pseudobulbar Affect (Involuntary Laughing and/or Crying)
Keywords: PBA; involuntary crying; involuntary laughing
MeSH Terms: interventions — dextromethorphan - quinidine combination; Dextromethorphan; Quinidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NUEDEXTA® (Other): NUEDEXTA capsules (20 mg dextromethorphan hydrobromide and 10 mg quinidine sulfate) administered orally, once a day from Days 1 to 7 and twice a day from Days 8 to 180
  Interventions: Drug: NUEDEXTA®

INTERVENTIONS:
Drug: NUEDEXTA® — NUEDEXTA® only
  Other Names: dextromethorphan hydrobromide and quinidine

SUMMARY:
6 month study of NUEDEXTA ® (Dextromethorphan Hydrobromide and Quinidine Sulfate) for the treatment of Pseudobulbar Affect (PBA) in Nursing Home Patients.

DETAILED DESCRIPTION:
Eligible patients for this study must have a diagnosis of a neurological disorder affecting the brain of at least 3 months duration prior to baseline and which is not rapidly progressing and must have a diagnosis of Pseudobulbar affect (PBA).

This is a multicenter, open label study consisting of 6 months of treatment.

Approximately 125 patients will be enrolled at approximately 25 centers in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a neurological disorder affecting the brain (e.g. Alzheimer's and other dementias, stroke, Trauma Brain Injury, Multiple Sclerosis, Amyotrophic Lateral Sclerosis, Huntington's disease, Parkinson's disease) of at least 3 months duration prior to baseline and which is not rapidly progressing
* Diagnosis of Pseudobulbar Affect (PBA)
* A Center for Neurologic Study-Lability Scale (CNS-LS) score of 13 or greater at Baseline
* Minimum Data Set (MDS) information for patient available within 60 days prior to Baseline
* Informant who is willing to comply with study procedures

Exclusion Criteria:

* Patients who have received NUEDEXTA® in the past 1 year
* Patients with the diagnosis of Severe Depressive Disorder that would interfere with the conduct of the study
* Patients who have a history of schizophrenia spectrum and other psychotic disorders
* Patients with co-existent clinically significant or unstable systemic diseased that could confound the interpretation of the safety results of the study (e.g.,malignancy, poorly controlled diabetes, poorly controlled hypertension, unstable pulmonary, renal or hepatic disease, unstable ischemic cardiac disease, dilated cardiomyopathy, or unstable valvular heart disease)
* Patients with myasthenia gravis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Miami, Florida
  - Centerville, Ohio

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 14 participants were screened for study enrollment; however, only 5 participants were enrolled.
Groups:
- 20 mg Dextromethorphan Hydrobromide/10 mg Quinidine Sulfate: Participants received 20 milligrams (mg) dextromethorphan hydrobromide/10 mg quinidine sulfate capsules administered orally, once a day from Day 1 to Day 7 and twice a day from Day 8 to Day 180.
Period: Overall Study
Arm/Group | 20 mg Dextromethorphan Hydrobromide/10 mg Quinidine Sulfate
Started | 5
Completed | 1
Not Completed | 4
Not completed — Adverse Event | 3
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | 20 mg Dextromethorphan Hydrobromide/10 mg Quinidine Sulfate
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Scores on the Center for Neurologic Study-Lability Scale (CNS-LS)
Description: The study was terminated prematurely because of difficulty with recruiting. Analysis for this outcome measure was not performed because data were not collected prior to termination.
Time Frame: 180 days
Arm/Group | 20 mg Dextromethorphan Hydrobromide/10 mg Quinidine Sulfate
Number analyzed (Participants) | 0

2. Primary Outcome: Scores on the Clinical Global Impression of Severity of Illness (CGIS) Scale
Description: as for outcome 1
Time Frame: 180 days
Arm/Group | 20 mg Dextromethorphan Hydrobromide/10 mg Quinidine Sulfate
Number analyzed (Participants) | 0

3. Primary Outcome: Scores on the Clinical Global Impression of Change (CGIC) Scale
Description: as for outcome 1
Time Frame: 180 days
Arm/Group | 20 mg Dextromethorphan Hydrobromide/10 mg Quinidine Sulfate
Number analyzed (Participants) | 0

4. Primary Outcome: Scores on the Patient Global Impression of Change (PGIC) Scale
Description: as for outcome 1
Time Frame: 180 days
Arm/Group | 20 mg Dextromethorphan Hydrobromide/10 mg Quinidine Sulfate
Number analyzed (Participants) | 0

5. Primary Outcome: Number of Participants With the Indicated Responses to the Neuropsychiatric Inventory-Nursing Home (NPI-NH) Questionnaire
Description: as for outcome 1
Time Frame: 180 days
Arm/Group | 20 mg Dextromethorphan Hydrobromide/10 mg Quinidine Sulfate
Number analyzed (Participants) | 0

6. Primary Outcome: Scores on the Impact of Pseudobulbar Affect (PBA) on Participant Scale
Description: as for outcome 1
Time Frame: 180 days
Arm/Group | 20 mg Dextromethorphan Hydrobromide/10 mg Quinidine Sulfate
Number analyzed (Participants) | 0

7. Primary Outcome: Scores on the Minimum Data Set (MDS) Sections of Presumed Relevance to PBA, Including Sections on Speech, Cognition, Mood, Behavior, Health Condition, and Medication
Description: as for outcome 1
Time Frame: 180 days
Arm/Group | 20 mg Dextromethorphan Hydrobromide/10 mg Quinidine Sulfate
Number analyzed (Participants) | 0

8. Primary Outcome: Number of Participants Using Concomitant Psychotropic Medication
Description: as for outcome 1
Time Frame: 180 days
Arm/Group | 20 mg Dextromethorphan Hydrobromide/10 mg Quinidine Sulfate
Number analyzed (Participants) | 0

9. Primary Outcome: Scores on the Impact of PBA on Informant Scale
Description: as for outcome 1
Time Frame: 180 days
Arm/Group | 20 mg Dextromethorphan Hydrobromide/10 mg Quinidine Sulfate
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | 20 mg Dextromethorphan Hydrobromide/10 mg Quinidine Sulfate
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 20 mg Dextromethorphan Hydrobromide/10 mg Quinidine Sulfate (N=5)
Altered mental status (Psychiatric disorders) | 1
Severe agitation (Psychiatric disorders) | 1
Worsening of urinary tract infection (Infections and infestations) | 1
Left leg tibia fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 20 mg Dextromethorphan Hydrobromide/10 mg Quinidine Sulfate (N=5)
Urinary tract infection (Infections and infestations) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1

LIMITATIONS AND CAVEATS:
The study was terminated prematurely because of difficulty with recruiting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other